CLINICAL TRIAL: NCT05194501
Title: EVALUATION OF THE FUNCTIONAL STATUS OF THE "UNAFFECTED" HAND IN HEMIPLEGIC PATIENTS
Brief Title: Unaffected Hand in Hemiplegia
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, Lecturer Doctor, Ufuk University
Other Study IDs: 2021-04-04
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Hemiplegia; Upper Extremity Problem
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nine Hole Peg Test, Jamar dynamometer, pinchmeter — Hand grip and pinch strengths: Hand grip strengths and tip pinch strengths were measured using a Jamar type hand dynamometer and pinchmeter available in our clinic.
  The Nine Hole Peg Test (NHPT): Hand dexerities were evaluated with the NHPT available in our clinic.

SUMMARY:
The primary aim of our study is to evaluate the functional status of the unaffected hand in hemiplegic patients. The secondary aims are to compare the functional states of the unaffected hand between right and left hemiplegias, and to evaluate the relationships between the functional status of the unaffected hand and the healing phase of the hemiplegic side and activities of daily living.

This cross-sectional study included 30 right hemiplegic and 30 left hemiplegic patients with a history of ischemic cerebrovascular accident (CVA) in the last 1 year and 30 healthy volunteers as a control group.

Participants' data on age, gender, height, weight, comorbidities, time after stroke, and affected body half were recorded. In the patient group, the stages for the upper extremity and hand were evaluated according to the Brunnstrom recovery stages. Afterwards, the participants' hand grip strengths were evaluated with a Jamar type hand dynamometer, pinch strengths with a pinchmeter, and hand dexerity with the Nine Hole Peg Test (NHPT). Evaluations were made in the unaffected hand in the patient groups and in both hands in the control group. The Lawton Instrumental Activities of Daily Living Scale (Lawton-IADL) and the Functional Independence Measure (FIM) were applied to the patient groups.

ELIGIBILITY:
Inclusion Criteria:

This cross-sectional study included 30 right hemiplegic and 30 left hemiplegic patients with a history of ischemic cerebrovascular accident (CVA) in the last 1 year and 30 healthy volunteers as a control group. All patients and healthy volunteers were right hand dominant.

Exclusion Criteria:

Patients with a history of CVA in the last 1 month, bilateral hemispheric ischemic lesion, moderate/severe cognitive impairment, aphasia, neglect, and patients/healthy volunteers with severe systemic, inflammatory, degenerative and neurological diseases that may lead to loss of hand functions, a history of surgery or trauma in the upper extremity in the last 3 months, and younger than 18 years of age were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study included 30 right hemiplegic and 30 left hemiplegic patients with a history of ischemic cerebrovascular accident (CVA) in the last 1 year and 30 healthy volunteers as a control group.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Hand grip and pinch strengths | 6 month
  Hand grip and pinch strengths: Hand grip strengths and tip pinch strengths were measured using a Jamar type hand dynamometer and pinchmeter available in our clinic. The measurement of hand grip strengths were made with shoulders in adduction and neutral rotation, elbows in 90 degrees flexion, forearms and wrists in neutral position. Tip pinch strengths were measured by squeezing the pinchmeter between the thumb and forefinger [12]. Participants were asked to take a deep breath and grasp with maximal force while exhaling. The measurements were repeated three times with an interval of five minutes, and the average of the values was taken as the basis for the analyses.
The Nine Hole Peg Test (NHPT) | 6 month
  The Nine Hole Peg Test (NHPT): Hand dexerities were evaluated with the NHPT available in our clinic. This test is an assembly consisting of a square platform and storage box. There are nine holes in the square-shaped area and nine cylinders suitable for these holes. The patients are asked to take the 9 cylinders one by one from the storage box as quickly as possible, place them into the holes, and place them back in the storage box one by one after all the cylinders have been placed. Meanwhile, the total time is measured in seconds with the chronometer. Less time indicates better hand dexterity.
The Lawton Instrumental Activities of Daily Living Scale (Lawton-IADL) | 6 month
  The Lawton Instrumental Activities of Daily Living Scale (Lawton-IADL): Lawton-IADL scale is a scale consisting of eight questions questioning activities use a phone, food preparation, shopping, housekeeping, laundry, use of public transportation, managing self-medication, and handling finances. Each question is scored as 0 (can not perform or can partially perform) or 1 (can perform) [5]. The total score ranges from 0 (low functionality, dependent) to 8 (high functionality, independent). The Turkish validity and reliability study of the scale was conducted by Işık et al. in 2020.
The Functional Independence Measure (FIM) | 6 month
  The Functional Independence Measure (FIM): FIM is an 18-item scale that evaluates the degree of independence of the individual in basic physical and cognitive activities in daily life. It has two main sections in which physical/motor function (13 questions) and cognitive function (5 questions) are evaluated. The part of physical/motor function consists of 4 sub-sections in which different activities [self-care performance (eating, grooming, bathing, upper dressing, lower dressing, toileting), sphincter control, transfers, locomotion] are evaluated. The part of cognitive function consists of 2 sub-sections in which communication and social-cognition are evaluated. Each item is scored from 1 to 7, with 'level 1' representing full assistance and 'level 7' being complete independence. The higher the total score, the higher the level of independence. The Turkish adaptation study of the scale was carried out in 2001 by Küçükdeveci et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided